CLINICAL TRIAL: NCT03855449
Title: Web-Based Problem Solving Self-Management Program for African Americans With Type 2 Diabetes
Brief Title: A Task Analysis Study of DECIDE For African American Patients With Type 2 Diabetes
Acronym: eDECIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Wichita State University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michelle Redmond, Assistant Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00141460; 1K01HL135472-01A1 (NIH)
Record Dates: First submitted 2019-02-20; First posted 2019-02-26 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Problem solving; Self-management; Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: A single group will be recruited to go through the in-person DECIDE problem-solving curriculum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eDECIDE Web-based Intervention Group (Experimental): Participants randomized to the eDECIDE arm will use the online version of the program through the eDECIDE study portal. Participants in this group will receive bi-weekly calls from their health coach to mark their progress with the program.
  Interventions: Behavioral: eDECIDE Web-based Intervention Group
- DECDIE Traditional Group (Active Comparator): Participants randomized to the DECIDE group will receive a copy of the curriculum via mail and will be a self-study group where they go through the curriculum on their own with 4 calls from their health coach.
  Interventions: Behavioral: eDECIDE Web-based Intervention Group

INTERVENTIONS:
Behavioral: eDECIDE Web-based Intervention Group — Will conduct 18 week in-person group sessions of the DECIDE curriculum with recruited volunteers. This is part 1 or phase I of the eventual pilot clinical trial. Participants will attend weekly group sessions to learn problem-solving skills and management of their diabetes.
  After the completion of the task analysis participants will be recruited for the eDECIDE web-based intervention

SUMMARY:
The Decision-Making Education for Choices in Diabetes Every Day (DECIDE) program (copyrighted) was created by Dr. Felicia Hill-Briggs and is used by permission for the purpose of this pilot study. This problem-solving curriculum is used to help manage everyday problems when living with diabetes. The purpose of this project is to complete an in-depth review of the Decision-Making Education for Choices in Diabetes Every Day (DECIDE) curriculum, which is delivered in a group face-to-face setting. Using a task analysis process, the investigators will use the findings from the review to develop a web-site version that will be called eDECIDE for use with a community group in Kansas.

Phase 2: will be a pilot clinical trial (2 Arm Study) which examines the use of the eDECIDE curriculum compared to the traditional DECIDE curriculum delivered to participants individually.

DETAILED DESCRIPTION:
The Task Analysis study of the DECIDE program is phase I (part 1) of a three-part study. Part 2 is usability testing and Part 3 is the pilot clinical trial. For part 1, a single group will receive the DECIDE intervention program as investigators conduct a task analysis of DECIDE in preparation for building the web-based version (eDECIDE). This web-based version will be used for part 3 of the study, which will be the pilot clinical trial (eDECIDE).

Self-management is important for persons with type 2 diabetes for glycemic control. When diabetes is uncontrolled, it is important to get back in control in order to decrease further health complications. New ways of delivering self-management that improve access to treatment are needed. This study will help provide background information on any potential problems and or benefit of using web-based and mobile phone applications (mHealth) for diabetes self-management. In addition, this study will help researchers at University of Kansas School of Medicine create a web-based version of the in-person DECIDE program, known as eDECIDE. Data gathered from the in-person DECIDE group sessions will be used to create a series of events for designing a web-based copy based on several task (current study). Therefore, this study is known as a task analysis.

Task Analysis: This entails documenting observations of an existing system, sequence of tasks, and information flows. High-level tasks are divided into subtasks and operations. Informational sources required in each subtask are also recorded. This technique is a critical step in any software development process to ensure a basic understanding of user needs and requirements necessary for optimal learning. It also provides a perspective on individual differences across patients. Understanding this workflow is critical and will serve as the basis for developing eDECIDE.

For the task analysis up to 8 individuals will be recruited to take part in the in-person DECIDE problem-solving curriculum (task analysis), the information learned in the task analysis will help build and test (usability testing) the eDECIDE website, which are both integral to the pilot clinical trial (part 3) which will take place last.

PROCEDURES The current study will administer the DECIDE curriculum to a single group, examine responses, build the website, and then prepare for implementing the pilot clinical trial. The information gathered from this study will provide information about barriers to problem solving for diabetes self-management and perceptions of using a web-based diabetes problem-solving format.

Participants who meet eligibility criteria will take part in 9-weekly sessions on diabetes self-management and problem-solving techniques. The sessions will be recorded by audio and video tape. All audio and video taped recordings will be used to help create the web-based version of DECIDE, known as eDECIDE. All and any personal information that is recorded by audio tape will be removed when transcribing the audio recordings. All personal information such as name and face will be removed and blurred if video recording clips are used in an academic or conference meeting setting. Other personal identifiable information such as date of birth, address, or telephone number will be removed when transcribing and you will be identified by participant id number. The researcher will ask participants questions about their diabetes self-management behaviors; go over problem-solving techniques, and self-management skills. The recordings of the focus group sessions will be destroyed 12 months after publication of the research results.

Task Analysis and usability testing Procedures:

Using information gathered from the task analysis, the research team will develop a wire frame prototype of eDECIDE. A benefit of the prototype is to have a layout of the interface without the distraction of color or visual elements that would normally be a part of the actual webpages.

Once the prototype of the website design is complete, investigators will conduct usability testing (part 2) to assess the efficiency, ease-of-use, and user satisfaction based on participant feedback. Participant feedback is collected via web camera and online questionnaires. Objective data are collected via logging software designed for usability testing. Usability testing is a step-by-step process conducted several times throughout the design and development process. Results from each test are used to make design recommendations for the eDECIDE website. Once usability testing is complete, the pilot clinical trial (part 3) of eDECIDE will begin.

Our long-term goal is to understand how problem-solving skills training (PSST), delivered using web-based and mobile phone technology, can improve diabetes self-management in community populations.

Currently Recruiting: Clinical Trial Phase of eDECIDE: Plot 2-Arm Study:

Intervention arm: eDECIDE Online Curriculum Comparison arm: DECIDE Traditional Curriculum delivered one/on/one (Self-Study).

Will recruit at total of 40-70 participants Primary outcome A1c Secondary outcomes: goal setting, problem-solving, feasibility of use for eDECIDE online, satisfaction with eDECIDE online.

ELIGIBILITY:
Inclusion Criteria:

* African American
* English speaking
* Access to the Internet daily
* Reading level of at least 5th grade
* Diagnosis of Type 2 Diabetes per one of the following

  1. Fasting blood glucose ≥ to 126 mg/dL
  2. 2 hr plasma glucose ≥ 200 mg/dL
  3. Glycosylated hemoglobin HbA1c ≥ to 6.5%
  4. Random plasma glucose ≥ 200 mg/dL

Exclusion Criteria:

* Glycosylated hemoglobin HbA1c ≤ 7.0
* Pregnancy
* Severe visual or hearing impairment or any existing condition that would limit or hinder one's ability to use the Internet
* Dementia
* Use of supplemental oxygen
* Chest pain or angina
* Prior lower extremity amputation
* A diagnosis of a life threatening malignancy within the past year

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Task Analysis study process chart | 15 weeks
  First output of the task analysis is a process chart of conducting the DECIDE program, using video tapped sessions of DECIDE
Task Analysis Wireframe Development part 1 | 15 weeks
  Second output of the task analysis is a task flow diagram of facilitation and participant responses using case scenarios by user group.
Task Analysis Wireframe Development part 2 | 15 weeks
  Third output of the task analysis is a task decomposition table of the DECIDE curriculum, breaking down the task/actions of facilitator and participant into smaller task for replicating on the website

CONTACTS AND LOCATIONS:
Overall Officials: Michelle L Redmond, PhD, Principal Investigator — University of Kansas Medican Center Research Institute, Inc
Locations (1):
- University of Kansas Medical Center, Wichita, Kansas, United States

IPD SHARING:
Plan to Share IPD: No